CLINICAL TRIAL: NCT05036421
Title: Effect of UGT Genetic Variation on Pharmacokinetics of Empagliflozin
Brief Title: Effect of Glucuronosyltransferase (UGT) Genetic Variation on Pharmacokinetics of Empagliflozin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHCL277
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Pharmacogenomic; Pharmacokinetics
Keywords: UGT polymorphism; Pharmacokinetics; Empagliflozin
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: open label, single-dose, one-period, design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Empagliflozin
  Interventions: Drug: Empagliflozin 10 milligram

INTERVENTIONS:
Drug: Empagliflozin 10 milligram — antihyperglycemic medication
  Other Names: Jardiance

SUMMARY:
The aim of this works is to investigate the effect of genetic polymorphism of snps on human response to treatment with empagliflozin and its correlation with with pharmacokinetic parameters in Egyptian subjects

DETAILED DESCRIPTION:
Empagliflozin is a sodium glucose co-transporter-2 (SGLT-2) inhibitor indicated as an adjunct to diet and exercise to improve glycemic control in adult patients with type 2 diabetes. SGLT2 co-transporters are responsible for reabsorption of glucose from the glomerular filtrate in the kidney. The glucuretic effect resulting from SGLT2 inhibition reduces renal absorption and lowers the renal threshold for glucose, therefore resulting in increased glucose excretion. Additionally, it contributes to reduced hyperglycaemia and also assists weight loss and blood pressure reduction.

ABSORPTION Following oral administration, peak plasma concentrations were reached at 1.5 hours post-dose and then declined in a biphasic manner with a rapid distribution phase and a relatively slow terminal phase. Administration following a high-fat and high-calorie meal results in a slightly lower exposure with area under the curve (AUC) decreasing by approximately 16% and Cmax decreasing by approximately 37% compared to fasted condition.

METABOLISM In vitro studies suggest that empagliflozin is primarily metabolized by glucuronidation by 5'-diphospho-glucuronosyltransferases UG2B7, UGT1A3, UGT1A8, and UGT1A9. The most abundant metabolites are three glucuronide metabolites: 2-O-, 3-O-, and 6-O-glucuronide. Empagliflozin does not inhibit, inactivate, or induce CYP450 isoforms. It is a substrate for p-glycoprotein (p-gp), however in vitro studies suggest that it is unlikely to cause interactions with drugs that are p-gp substrates.

After oral administration, empagliflozin was 41.2% eliminated in feces and 54.4% eliminated in urine.

Terminal elimination half life was found to be 12.4 h based on population pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers
* Age between (18-45 years)
* Normal BMI.
* Understand the procedures and are willing to participate and gave their final written consent prior to the commencement of the study procedures.
* The volunteers will be asked to provide a complete medical history, and complete a physical examination, laboratory tests [hematology, clinical chemistry, urinalysis, serology (including hepatitis B surface antigen, anti-hepatitis C virus and antihuman immunodeficiency virus antibody).

Exclusion Criteria:

* Treatment with any known enzyme-inducing/inhibiting agents within 30 days prior to the start of the study and throughout the study.
* Subjects who have taken any medication less than two weeks of the trials starting date.
* Susceptibility to allergic reactions to study drugs.
* Any prior surgery of the gastrointestinal tract that may interfere with drug absorption.
* Gastrointestinal diseases.
* Renal diseases.
* Cardiovascular diseases.
* Pancreatic disease including diabetes.
* Hepatic diseases.
* Hematological disease or pulmonary disease
* Abnormal laboratory values.
* Subjects who have donated blood or who have been involved in multiple dosing study requiring a large volume of blood (more than 500 ml) to be drawn within 6 weeks preceding the start of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 48 hours
  AUC0→∞
Bioavailability parameters | 24 hours
  Cmax

SECONDARY OUTCOMES:
Secondary outcome | 48 hours
  Tmax

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Shaheen, Assiss. Prof, Principal Investigator — Ain Shams University
Locations (1):
- Faculty of Pharmacy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No